CLINICAL TRIAL: NCT04939103
Title: TRUS-FNA Versus MRI， CT， Enteroscopy, Superficial Biopsy, TRUS For The Prediction Of pCR After Neoadjuvant Treatment In Rectal Cancer
Brief Title: TRUS-FNA For The Prediction Of pCR After Neoadjuvant Treatment In Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Chief Physician, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: luoyanxin
Record Dates: First submitted 2021-06-03; First posted 2021-06-25 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: EUS-FNA; Rectal Cancer; Pathological Complete Remission
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- 1: Those patients with rectal cancer after neoadjuvant treatment and completed the examination of TRUS-FNA, TRUS, CT, MR, enteroscopy and superficial biopsy
  Interventions: Device: TRUS-FNA

INTERVENTIONS:
Device: TRUS-FNA — Transrectal Ultrasound Guided Fine Needle Aspiration for rectal tumor

SUMMARY:
Colorectal cancer is one of the most malignancies worldwide. The dominant clinical research strategy of LARC includes neoadjuvant chemoradiotherapy before radical surgery followed combined with adjuvant treatment. Approximately 15% to 20% of the patients after nCRT can achieve a pathologic complete response (pCR)---no residual tumor is reported at histology after a standard resection. Some researchers suggest that those patients with pCR can be spared the morbidities of surgery instead by a nonoperative approach---watch- and-wait(W&W). However, neither FDG-PET, MRI, CT, nor enteroscopy can accurately determine a pCR.

EUS-FNA has been an important technique for the diagnosis of rectal cancer for its high accuracy and little harm. However, data on the TRUS-FNA for the cytologic diagnosis of pCR in rectal cancer is scarce. Our hypothesis is that adding transrectal ultrasound-guided fine needle aspiration (TRUS-FNA) compared with enteroscopy , MR, and CT alone can improve the accuracy of predicting pCR after nCRT.Therefore, the aim of the study is to assess the performance characteristics of EUS-FNA in this setting.

DETAILED DESCRIPTION:
Following the neoadjuvant treatment of rectal cancer, appropriately 15-20%of patients receiving neoadjuvant treatment can achieve pathological complete response: a condition of no tumor cell detected in surgical specimens, which usually suggests improved oncology outcomes. In 2004, Habr-Gama, A et al. proposed that surgical resection may not increase overall and disease-free survival in these patients and lead to an increased risk of surgical complications and permanent stoma. Therefore, they suggested that nonoperative treatment, which is now referred to as "watch-and-wait"--patients with clinical complete response (cCR) can avoid unnecessary surgery and be managed by strict follow-up and observation alone. A series of studies have shown impressive survival outcomes in patients who received nonoperativetreatment:85-93% and 82-94% in 5-year overall survival and disease-free survival, respectively. Also, in case of relapse, the rate of successfully performed salvage surgery was 80-91%.

However, determining pCR after neoadjuvant treatment for distal rectal cancer remains a dilemma for clinicians. Different imaging modalities, including digital rectal examination (DRE), fludeoxyglucose positron emission tomography (FDG-PET), Computed Tomography (CT), magnetic resonance imaging (MRI), transrectal ultrasound (TRUS) and endoscopy have been well evaluated for the efficacy of predicting pCR. In contrast, none of them proved to be reliable.

Duldulao et al. found that after neoadjuvant treatment, rectal tumor cells are distributed preferentially in the muscularis of the bowel wall while few in the mucosa. That is why superficial biopsies were inadequate, and full-thickness apparitions on tumor focus may provide adequate sampling to rule out malignancy for all stages of rectal cancer after neoadjuvant treatment. Therefore, fine-needle aspiration assisted with TRUS (TRUS-FNA), which can harvest a whole layer of the bowel wall, has shown obvious advantages in this setting.

Although widely used in clinical practice, studies regarding the application of TRUS-FNA in predicting pCR after preoperative therapy of rectal cancer were scarce. We hypothesized that TRUS-FNA could improve the clinical practice of identifying patients achieving pCR after neoadjuvant treatment. Accordingly, we conducted this prospective study to evaluate the efficacy of TURS-FNA, compared with other imaging modalities, TRUS, MRI, CT, enteroscopy, and superficial biopsy, in predicting pCR of rectal cancer after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* a new diagnosis of histologically confirmed rectal adenocarcinoma
* tumor located below the peritoneum reflex
* over 18 years old
* T1-4,N0-2,M0 before nCRT
* complete nCRT treatment
* ASA>III or ECOG>1
* informed consent

Exclusion Criteria:

* multiple primary colorectal cancer
* the history of malignant tumor,IBD,FAP
* the history of chemoradiation treatment or resection of rectal tumor
* actue abdomen disease requiring emergency surgery
* not be able to tolerate surgery with severe organ dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all of the patients are from the sixth affiliated hospital of Sun Yet-sen University
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
the accuracy of predicting pCR after nCRT | 25/05/2021-25/05/2022
  The primary endpoint was the predictive yield of TRUS-FNA for pathological complete responses after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: luo yanxin, MD,PHD, Study Chair — the sixth affiliated hospital of Sun Yet-Sen University
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.